CLINICAL TRIAL: NCT03489759
Title: The Effect of Vitamin E-coated Polysulfone Membrane on Oxidative Stress, Inflammation and Monocytes in Critically Ill Patients in CRRT: a Pilot, Randomized, Double-blinded, No-profit, Clinical Study
Brief Title: The Effect of Vitamin E-coated Polysulfone Membrane on Oxidative Stress, Inflammation and Monocytes in Critically Ill Patients in CRRT
Acronym: Vitabrane E
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: St. Bortolo Hospital (Other)
Responsible Party: Principal Investigator, Silvia De Rosa, Medical Doctor, St. Bortolo Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 79/16A
Record Dates: First submitted 2018-03-13; First posted 2018-04-05 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: Renal Failure; Renal Insufficiency, Acute
Keywords: Acute Kidney Injury; Oxidative Stress; Renal Replacement Therapy; Vitamine E-coated Polysulfone Membrane
MeSH Terms: conditions — Renal Insufficiency; Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The randomization list will be kept in a special lockable closet, not accessible to the other investigators involved in the study. The one who will create the list will not be involved in any other role in the present study.
  The filter label, and hence the name, will be covered by a white covering label. Each kit of filters needed to perform a single treatment will be prepared in a closed box and the patient number will be written on it, so that the user who performs the treatment will not be able to understand which filter it is.
  All the other investigators involved in the present study (nurses in the Nephrology department who will follow the treatment, the researchers who will collect the clinical data, the biologists who will analyze the samples and the statisticians who will analyze the data) will not know which filter has been applied in each treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ViE15-A (Experimental): The patients were randomly allocated to two groups by using computer-generated numbers. The renal replacement therapy will be started using ViE15-A hemofilter
  Interventions: Device: ViE15-A
- REXEED-15A (Active Comparator): TThe patients were randomly allocated to two groups by using computer-generated numbers. The renal replacement therapy will be started using REXEED-15A
  Interventions: Device: REXEED-15A

INTERVENTIONS:
Device: ViE15-A — The type of dialytic treatment that will be used during the study will be continuous venous hemofiltration (CVVH-Continuous veno-venous hemofiltration). The filter will be ViE15-A.
  Arms: ViE15-A
Device: REXEED-15A — The type of dialytic treatment that will be used during the study will be continuous venous hemofiltration (CVVH-Continuous veno-venous hemofiltration). The filter will be REXEED-15A.
  Arms: REXEED-15A

SUMMARY:
The study evaluate the effect of a membrane in polysulfone covered with vitamin E (ViE15-A, ASAHI Kasey, Tokyo, Japan) versus non-vitamin E polysulfone membrane (REXEED-15A, ASAHI Kasey, Tokyo, Japan) in critically ill patients admitted to intensive care undergoing continuous extracorporeal dialysis (CRRT).

The current randomized study is designed to assess the effect on the levels of oxidative stress, pro and anti-inflammatory cytokines and the mode and amount of death of monocytic cell lines using ViE 15-A in comparison withe REXEED-15A.

The investigators hypothezise that the ViE15-A versus REXEED-15A will have different effect on the levels of oxidative stress, pro and anti-inflammatory cytokines and the mode and amount of death of monocytic cell lines.

DETAILED DESCRIPTION:
The study evaluate the effect of a membrane in polysulfone covered with vitamin E (ViE15-A, ASAHI Kasey, Tokyo, Japan) on the levels of oxidative stress, pro and anti-inflammatory cytokines and the mode and amount of death of monocytic cell lines in critically ill patients admitted to intensive care undergoing continuous extracorporeal dialysis (CRRT).

This membrane will be compared with a non-vitamin E polysulfone membrane (REXEED-15A, ASAHI Kasey, Tokyo, Japan) and already intended for use in continuous renal support therapy.

The current randomized study is designed to assess the effect on the levels of oxidative stress, pro and anti-inflammatory cytokines and the mode and amount of death of monocytic cell lines using ViE 15-A in comparison withe REXEED-15A.

Precisely, will be evaluated

1. the effect of the filter on the reduction of the plasma levels of two pro-inflammatory cytokines (IL-1β and IL-6) and of two anti-inflammatory cytokines (IL-10, IL-8);
2. the analysis of the life modality of the monocytic cells: the patient's plasma will be used, incubated for 24 hours with U937 cells (monocyte precursor cells), necrosis cells and the percentage of apoptotic cells. The apoptotic cells will also evaluate the apoptotic pathway (evaluation of activated caspases) that led to cell death. The differences that are highlighted in the two different sampling moments become expressed Δ% with respect to the initial value Secondary outcomes will be to evaluate the clinical outcomes (haemodynamic and hematochemical parameters) in the short and long term deriving from the application of a membrane with vitamin E; for this reason, for the whole duration of the extracorporeal dialysis therapy, the same filter assigned to the patient at the time of enrollment will be used.

All the other parameters of the extracorporeal treatment that can influence the results will be standardized; in particular, the flows will be fixed according to the dialysis dose criteria and re-infusion methods according to the table in the paragraph "treatment characteristics".

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Acute Kidney Injury
* ICU patients with clinical indication for Continuous Renal Replacement Therapy
* Clinical decision to begin CVVH for at least 24 hours with high flux filter (defined as membranes with an ultrafiltration coefficient KUF > 25ml/Kg/h)
* Obtain the informed consent

Exclusion Criteria:

* Hemodialysis patients, peritoneal dialysis patients and transplant recipient;
* Hypothermia (T < 36°C)
* Regional Anticoagulation with Citrate
* Septic Shock;
* Neoplasm in Chemotherapy
* Extra-Corporeal Membrane Oxygenation
* Cardio Circulatory Arrest
* Autoimmune disease or immunosuppressed patients;
* Life expectancy < 24 hr
* Pregnancy;
* Informed Consent refused by the patient or surrogate decision-maker

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-03-13 (Actual); Primary Completion 2018-09-13 (Actual); Study Completion 2019-12-13 (Estimated)

PRIMARY OUTCOMES:
Copper/Zinc | change from 24 to 72 hours
  In vivo comparison of ROS concentrations in two groups
Superoxide Dismutas | change from 24 to 72 hours
  In vivo comparison of ROS concentrations in two groups
Endogenous peroxidase activity | change from 24 to 72 hours
  In vivo comparison of ROS concentrations in two groups
Nitric Oxide | change from 24 to 72 hours
  In vivo comparison of ROS concentrations in two groups
Viability | change from 24 to 72 hours
  Ex vivo comparison of relative decrease of monocytes cell line incubated in plasma
Apoptosis | change from 24 to 72 hours
  Ex vivo comparison of relative decrease of monocytes cell line incubated in plasma
Necrosis | change from 24 to 72 hours
  Ex vivo comparison of relative decrease of monocytes cell line incubated in plasma
Interleukine-6 | change from 24 to 72 hours
  In vivo comparison of relative reductions of inflammatory cytokines concentrations in two groups
Interleukine -10 | change from 24 to 72 hours
  In vivo comparison of relative reductions of inflammatory cytokines concentrations in two groups
Interleukine-18 | change from 24 to 72 hours
  In vivo comparison of relative reductions of inflammatory cytokines concentrations in two groups

SECONDARY OUTCOMES:
Comparison of CRRT-free days from enrollment to ICU discharge in two groups | 7 days
  The assessment of the effect of both hemofilters on short term clinical renal outcomes
Comparison of mechanical Ventilation-free days from enrollment to ICU discharge in two groups | 7 days
  The assessment of the effect of both hemofilters on short term clinical renal outcomes
Comparison of vasopressor drugs-free days in two groups | 7 days
  The assessment of the effect of both hemofilters on short term clinical renal outcomes
Comparison of ICU length of stay in two groups | 7 days
  The assessment of the effect of both hemofilters on short term clinical renal outcomes
Comparison of renal recovery in two groups | 7 days
  The assessment of the effect of both hemofilters on short term clinical renal outcomes
Comparison of CRRT-free days from enrollment to hospital discharge in two groups | 90 days
  The assessment of the effect of both hemofiltes on long term clinical renal outcomes
Comparison of need of (Intermittent Hemodialysis) IHD at hospital discarge in patients treated with vitamine E-coated membrane and non-vitamin E-coated membrane | 90 days
  The assessment of the effect of both hemofiltes on long term clinical renal outcomes
Comparison of renal recovery at hospital discharge in two groups | 90 days
  The assessment of the effect of both hemofiltes on long term clinical renal outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Ronco, MD, Study Director — Department of Nephrology, Dialysis and Transplantation
Locations (1):
- San Bortolo Hospital, Vicenza, Italy